CLINICAL TRIAL: NCT01623622
Title: A Phase 2 Study of HC-58 in Patients With Severe Upper Limb Hemiplegia After Stroke
Brief Title: Study of HC-58 in Upper Limb Hemiplegic Patients After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HC-58 (SHS) II-1
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2015-02

CONDITIONS: Severe Upper Limb Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HC-58 low dose (Experimental): Low dose
  Interventions: Drug: HC-58
- HC-58 high dose (Experimental): High dose
  Interventions: Drug: HC-58
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HC-58 — once or more / week
  Arms: HC-58 high dose; HC-58 low dose
Drug: Placebo — once or more / week
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of HC-58 in patients with severe upper limb hemiplegia following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe upper limb hemiplegia after stroke
* Within 28 days after stroke at enrollment

Exclusion Criteria:

* Patients with sensory loss between shoulder and hand on paralyzed side
* Patients with pain between shoulder and hand on paralysed side which affects medical rehabilitation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Onset of shoulder hand syndrome | 12 weeks
  The incidence rate of shoulder hand syndrome
Change from Baseline in the modified Barthel index (MBI) and MBI efficiency | 12 weeks
  MBI efficiency means MBI gain divided by period of administration
Change from Baseline in the Fugl-Meyer Assessment (FMA) (upper limb) and FMA efficiency | 12 weeks
  FMA efficiency means FMA gain divided by period of administration

SECONDARY OUTCOMES:
Pain score by numeric rating scale | 12 weeks
Swelling asymmetry between hands | 12 weeks
Discolouration of the skin of the hand | 12 weeks
Difference in skin temperature between hands | 12 weeks
Decreased range of motion | 12 weeks
Radiographic finding of bone | 12 weeks
Bone metabolic marker | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshiya Umeda, Study Director — Asahi Kasei Pharma Corporation Clinical Development Center
Locations (3):
- Japan (3):
  - Fukui-shi, Fukui
  - Hamamatsu, Shizuoka
  - Kumamoto, Kumamoto